CLINICAL TRIAL: NCT00957931
Title: Pilot Study MUD HCT:Pts High Risk Sickle Cell,Other Non-Malignant RBC Disorders- Reduced Intensity Preparative Regimen, HAPLO-Identical Mesenchymal Stromal Cells
Brief Title: Allo-HCT MUD for Non-malignant Red Blood Cell (RBC) Disorders: Sickle Cell, Thal, and DBA: Reduced Intensity Conditioning, Co-tx MSCs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Minnesota (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sandhya Kharbanda, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC01
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Sickle Cell Disease; Thalassemia; Diamond-Blackfan Anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Anemia, Diamond-Blackfan | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal stromal cells (Experimental)
  Interventions: Procedure: Bone marrow transplantation; Biological: Mesenchymal Stromal Cells

INTERVENTIONS:
Procedure: Bone marrow transplantation — Bone marrow transplantation using matched unrelated donors, reduced intensity conditioning regimen, and co-transplanting mesenchymal stromal cells derived from parental bone marrow.
Biological: Mesenchymal Stromal Cells

SUMMARY:
The main purpose of this project is to cure patients with high risk Sickle cell disease and other red cell disorders including thalassemia and diamond-blackfan anemia by bone marrow transplantation. The patients enrolled in this study will be those who lack matched sibling donors and therefore have no other option but to undergo bone marrow transplantation using matched but unrelated bone marrow or umbilical cord blood from the national marrow donor program registry. Since bone marrow transplantation for these disorders using matched unrelated donors has two major problems i.e. engraftment, or , the process of new marrow being accepted and allowed to grow in the the patient; and graft-versus-host disease, or the process where the new marrow "rejects" the host or the patient, this study has been devised with methods to overcome these two problems and thus make transplantation from unrelated donors both successful in terms of engraftment and safe in terms of side effects, both acute and long term.

In order to accomplish these two goals, two important things will be done. Firstly, patients will get three medicines which are considered reduced intensity because they are not known to cause the serious organ damage seen with conventional chemotherapy. These medicines, however, do cause intense immune suppression so these can cause increased infections. Secondly, in addition to transplantation of bone marrow from unrelated donors, patients will also transplanted with mesenchymal stromal cells derived from the bone marrow of their parents. Mesenchymal stromal cells are adult stem cells that are normally found in the bone marrow and are thought to create the right background for the blood cells to grow. They have been shown in many animal and human studies to improve engraftment. In addition, they have a special property by which they prevent and are now even considered to treat graft versus host disease. Therefore, by using a reduced intensity chemotherapy regimen before transplant and transplanting mesenchymal stromal cells, we hope to improve engraftment while at the same time decrease the potential for severe side effects associated with a conventional transplant which uses extremely high doses of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease (SCD) 1-25 years of age with an HLA-identical, but unrelated, donor or 1 human leukocyte antigen (HLA) allele mismatched bone marrow or up to 2 HLA antigen mismatched umbilical cord blood (UCB) donor with one or more of the following:

  * Stroke, central nervous system (CNS) hemorrhage or a neurologic event lasting longer than 24 hours.
  * Acute chest syndrome with a history of recurrent hospitalizations or exchange transfusions.
  * Recurrent vaso-occlusive pain, 3 or more episodes per year for 3 years or more years; or recurrent priapism.
  * Impaired neuropsychological function and/or abnormal cerebral MRI scan or abnormal transcranial Doppler (TCD).
  * Stage I or II sickle lung disease.
  * Sickle nephropathy (moderate or severe proteinuria or a glomerular filtration rate (GFR) 30-50% of the predicted normal value).
  * Bilateral proliferative retinopathy and major visual impairment in at least one eye.
  * Osteonecrosis of multiple joints with documented destructive changes.
  * Requirement for chronic transfusions but with RBC alloimmunization >2 antibodies during long term transfusion therapy.
  * Failure of hydroxyurea (HU) therapy.
* Patients aged 0-21 years with transfusion dependent alpha- or beta-thalassemia who have an HLA-identical or 1 HLA allele mismatched bone marrow or up to 2 HLA mismatched UCB donor.
* Patients aged 0-21 years with Diamond-Blackfan anemia who have an HLA-identical or 1 HLA allele mismatched bone marrow or up to 2 HLA mismatched UCB donor. Diamond- Blackfan anemia patients will only be eligible if they have failed steroid therapy.

Exclusion Criteria:

* Patients with one or more of the following:

  * Karnofsky or Lansky performance score <70 (See Appendices I and II).
  * Stage III-IV lung disease (Appendix III).
  * GFR<30% predicted normal values.
  * Pregnant or lactating females.
  * Active serious infection whereby patient has been on intravenous antibiotics for one week prior to study entry.
  * Any patient with AIDS or HIV seropositivity.
  * Any patient with invasive aspergillus infection within one year of study entry.
  * Psychologically incapable of undergoing bone marrow transplant (BMT) with associated strict isolation or documented history of medical non-compliance.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Kharbanda, M.D., Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Result] Kharbanda S, Smith AR, Hutchinson SK, McKenna DH, Ball JB, Lamb LS Jr, Agarwal R, Weinberg KI, Wagner JE Jr. Unrelated donor allogeneic hematopoietic stem cell transplantation for patients with hemoglobinopathies using a reduced-intensity conditioning regimen and third-party mesenchymal stromal cells. Biol Blood Marrow Transplant. 2014 Apr;20(4):581-6. doi: 10.1016/j.bbmt.2013.12.564. Epub 2013 Dec 24. PMID 24370862

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesenchymal Stromal Cells: Patients received bone marrow transplantation using matched unrelated donors, reduced intensity conditioning regimen, and co-transplanting mesenchymal stromal cells derived from parental bone marrow.
Period: Overall Study
Arm/Group | Mesenchymal Stromal Cells
Started | 6
Completed | 2
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 10 [8 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Number of known transfusions prior to HSCT [Median (Full Range); unit: transfusions] — HSCT = hematopoietic stem cell transplantation
  transfusions | 47.5 [4 to 220]
Diagnosis [Count of Participants; unit: Participants]
  Sickle cell disease | 4
  Thalassemia major | 2

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Stable Engraftment Post Hematopoietic Cell Transplantation (HCT)
Description: Stable engraftment was defined as absolute neutrophil count (ANC) >500 cells /µL for 3 consecutive days and platelet count >50,000 for one week without transfusion; subsequently stable engraftment was measured by percentage of donor cells.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 6
Participants | 3

2. Secondary Outcome: Overall Survival 6 Months Following HCT
Description: Overall survival is reported at the count of participants alive 6 months following HCT.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 6
Participants | 2

3. Secondary Outcome: Overall Survival 1 Year Following HCT
Description: Overall survival is reported at the count of participants alive 1 year following HCT.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 6
Participants | 2

4. Secondary Outcome: Count of Participants With Disease-free Survival 6 Months Following HCT
Description: Disease-free survival is defined as alive without underlying disease.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 6
Participants | 0

5. Secondary Outcome: Count of Participants With Disease-free Survival 1 Year Following HCT
Description: Disease-free survival is defined as alive without underlying disease.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Mesenchymal Stromal Cells
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mesenchymal Stromal Cells (N=6)
Graft failure with autologous recovery (Blood and lymphatic system disorders) | 2
SOS (Hepatobiliary disorders) | 1 — SOS = Sinusoidal obstruction syndrome
EBV-PTLD (Immune system disorders) | 1 — EPV = Epstein-Barr virus post-transplant lymphoproliferative disorder
Grade II GVHD (Immune system disorders) | 1 — GVHD = Graft-versus-host disease
Grade III acute GVHD (Immune system disorders) | 1
Adenovirus reactivation (Infections and infestations) | 1
BK virus reactivation (Infections and infestations) | 1
CMV pneumonitis (Infections and infestations) | 1 — CMV = Cytomegalovirus
CMV reactivation (Infections and infestations) | 1
CMV viremia (Infections and infestations) | 2
Disseminated toxoplasmosis (Infections and infestations) | 1
Gram-negative septic shock (Infections and infestations) | 1
HHV-6 viremia (Infections and infestations) | 1 — HHV-6 = Human Herpesvirus 6
Klebsiella and enterobacter (Infections and infestations) | 1
Klebsiella bacteremia (Infections and infestations) | 1
Intracranial bleeding (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
PRES (Nervous system disorders) | 1 — PRES = Posterior reversible encephalopathy syndrome

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes